CLINICAL TRIAL: NCT07392034
Title: Efficacy of Tranexamic Acid Reducing Blood Loss During Maxillofacial Trauma Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Shakir Hussain, Postgraduate resident Oral and maxillofacial surgery, Nishtar Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12076/NID
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hemoglobin Level Measurement; Blood Loss During Surgery; Duration of Surgery
Keywords: Tranexamic acid; Oral and maxillofacial trauma surgery; Blood loss; Hemoglobin; Duration of surgery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trenexamic acid group (Active Comparator): Thirty minutes prior to surgery, the intervention group received intravenous trenexamic acid at a dose of 20 mg/kg.
  Interventions: Drug: Tranexamic Acid (TXA)
- Placebo group (Placebo Comparator): Thirty minutes prior to surgery, the placebo group received 20 mL of normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Thirty minutes prior to surgery, the intervention group receive intravenous , single dose of tranexamic acid of 20 mg/kg.
  Arms: Trenexamic acid group
Drug: Normal saline — Thirty minutes prior to surgery, the placebo group received single dose of 20 mL of normal saline.
  Arms: Placebo group

SUMMARY:
Tranexamic acid (TXA) is an inexpensive, easily used and relatively safe drug. It inhibits plasminogen activation and plasmin thus retards clot disintegration.Therapeutic application of tranexamic acid in trauma for preventing blood loss has been documented since long. Since blood loss causes several serious complications, it is compensated emergently by transfusion of blood or its products. However, transfusion of blood and products always carries a risk of inadvertent transmission of infection, antigen-antibody reactions and additional cost all of which can be prevented if blood loss is reduced. Morbidity associated with the delay in compensating the blood loss could also be prevented by pharmaceutically preventing hemorrhage.

DETAILED DESCRIPTION:
During management of maxillofacial injuries, hemostasis is essential to clear the airway also. It is reported that blood loss is the most common complication following maxillofacial fractures and their treatment.TXA oral rinse has been used for preventing excessive hemorrhage for patients with coagulopathies. IV TXA has also been proven to be effective in reducing bleeding in healthy adults undergoing third molar surgery. Administration of TXA has also been evaluated and found effective in reducing post-surgical hemorrhage during and after bimaxillary orthognathic surgery.

This study has been planned to evaluate how efficacious is preoperative tranexamic acid in decreasing blood loss while performing surgery in cases with maxillofacial trauma in our local setting. the study results will provide local evidence and will support the incorporation of safe and inexpensive drug i.e., TXA into trauma clinical practice guidelines and local treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* either gender.
* presenting within seven days of trauma.
* planned for maxillofacial surgery.

Exclusion Criteria:

* Patients with international normalized ratio (INR) greater than 1.5.
* American Society of Anesthesiologists (ASA) physical status of 3 or higher.
* chronic kidney disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
mean intraoperative blood loss | Immediately at the end of surgery
  mean intraoperative blood loss between patients receiving intravenous tranexamic acid and those receiving placebo during maxillofacial trauma surgery.

SECONDARY OUTCOMES:
mean drop in hemoglobin levels postoperatively | 03 hours after post operatively
  To assess the mean drop in hemoglobin levels postoperatively between the TXA and placebo groups.
intraoperative blood transfusion | Preoperative
  To evaluate the need for intraoperative blood transfusion between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Saima Munir, FCPS (OMFS), Study Director — Nishtar institute of dentistry, Multan
Locations (1):
- Nishtar institute of dentistry, Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wong J, George RB, Hanley CM, Saliba C, Yee DA, Jerath A. Tranexamic acid: current use in obstetrics, major orthopedic, and trauma surgery. Can J Anaesth. 2021;68(6):894-917.
- [Background] Ramirez RJ, Spinella PC, Bochicchio GV. Tranexamic Acid Update in Trauma. Crit Care Clin. 2017;33(1):85-99.
- [Background] Patel PA, Wyrobek JA, Butwick AJ, Pivalizza EG, Hare GMT, Mazer CD, et al. Update on Applications and Limitations of Perioperative Tranexamic Acid. Anesth Analg. 2022;135(3):460-73.
- [Background] Gruen RL, Mitra B, Bernard SA, McArthur CJ, Burns B, Gantner DC, et al. Prehospital Tranexamic Acid for Severe Trauma. N Engl J Med. 2023;389(2):127-36.
- [Background] Colomina MJ, Contreras L, Guilabert P, Koo M, E MN, Sabate A. Clinical use of tranexamic acid: evidences and controversies. Braz J Anesthesiol. 2022;72(6):795-812.
- [Background] Wu B, Lv K. Effect of tranexamic acid on postoperative blood loss. Br J Oral Maxillofac Surg. 2024;62(5):489-92.
- [Background] Ockerman A, Vanassche T, Garip M, Vandenbriele C, Engelen MM, Martens J, et al. Tranexamic acid for the prevention and treatment of bleeding in surgery, trauma and bleeding disorders: a narrative review. Thromb J. 2021;19(1):54.
- [Background] Khiabani K, Ahmadfar M, Labafchi A, Gosheh MR, Samieirad S. Is Preoperative Administration of Tranexamic Acid Effective on Blood Loss Reduction in Mandibular Fracture Surgeries? A Triple-Blind Randomized Clinical Trial. J Oral Maxillofac Surg. 2021;79(2):429.e1-.e7.
- [Background] Dunphy L, Williams R. Immune thrombocytopenic purpura presenting with spontaneous gingival haemorrhage in pregnancy. BMJ Case Rep. 2019;12(1).
- [Background] Chen MWJ, Yong CW, Lum JL. Use of an improvised clamp to manage bleeding tongue injuries. Am J Emerg Med. 2021;39:252.e1-.e2.